CLINICAL TRIAL: NCT07208916
Title: Evaluation of Grape Consumption to Improve Muscle Strength and Cognitive Function
Brief Title: Evaluation of the Potential of Grape Consumption to Improve Muscle Strength and Cognitive Function
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Western New England University (Other)
Responsible Party: Principal Investigator, Brittany Adams, Associate Professor, Western New England University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: WNEIRB001
Record Dates: First submitted 2025-09-22; First posted 2025-10-06 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-10

CONDITIONS: Healthy
Keywords: grapes; diet; muscle strength; cognition; sarcopenia; serum biomarkers; women
MeSH Terms: conditions — Sarcopenia | interventions — whole grape extract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Grape Powder Arm (Experimental): All subjects will consume two 36g packets of grape powder (mixed with water) daily for two, 2-week periods during the study.
  Interventions: Dietary Supplement: Grape Powder

INTERVENTIONS:
Dietary Supplement: Grape Powder — All participants will consume two 36g packets of grape powder (mixed with water) daily for two, 2-week periods during the study. Participants will mix pre-measured grape powder with water and drink twice a day (once in the morning and in the afternoon/evening) for two weeks.

SUMMARY:
The goal of this clinical trial is to learn if eating grapes can improve muscle strength and thinking in generally healthy women over 65. The main questions it aims to answer are:

Does eating grapes improve muscle strength in women over 65? Does eating grapes improve cognition in women over 65?

Participants will be asked to take part in 4 sessions on campus. Each session will include:

Functional muscle strength testing Cognitive testing Blood draws

DETAILED DESCRIPTION:
The goal of this project is to perform a translational study to evaluate the potential of grape consumption to improve muscle and cognitive function with female human volunteers. The study will examine the impact of grape consumption on the functional strength and cognition of females over the age of 65. We will recruit 35 women who are in good overall health. On Day 1, consented participants will undergo baseline screening and assessments and will receive education on dietary restrictions for the following two weeks. After the two-week run-in diet period, on Day 14 participants will complete functional strength and cognitive testing, provide blood samples, and receive pouches of grape powder to be ingested daily. During the grape consumption phase of the trial, participants will ingest two 36 g pouches of grape powder daily for 30 days - equivalent to three servings of fresh grapes per day. Additional blood work, strength and cognitive testing will be performed on Day 28 and again on Day 42. Results will help to inform future studies on the effectiveness of regular grape intake on functional muscle strength and cognition in women over the age of 65, along with serum markers that are indicative of underlying mechanisms of action.

ELIGIBILITY:
Inclusion Criteria:

* Healthy female (confirmed by medical history)
* Aged 65 or older;
* Able to walk household distances without assistance from another person
* Non-smoker;
* Dominant hand grip strength at or below normal value for age and gender;
* Had not consumed recreational drugs for one week prior;
* Agreed not to participate in any clinical or patch test studies at Day 1 through study completion;
* Completed a medical intake;
* Read, understood, and signed an informed consent.

Exclusion Criteria:

* Using nasally inhaled/systemic/topical corticosteroids within 4 weeks prior to and/or during the study, or systemic/topical antihistamines 72 hours prior to and during the study;
* Using certain antifungal drugs, antihistamines (including diphenhydramine, or Benadryl), antibiotics 4 (including "sulfa" drugs, quinolones and tetracyclines), oral diabetes drugs, sulfonylureas, diuretics, and tricyclic antidepressants. Some herbal supplements such as St. John's Wort would make a person ineligible;
* Not willing to refrain from using acetaminophen (occasional use permitted, except within 48 hours of a study visit) or systemic/topical anti-inflammatory analgesics such as aspirin, Aleve, Motrin, Advil, Orudis, or Nuprin for 72 hours prior to and during study visits;
* Any of the following in the 4 weeks prior to start of study:

  1. Major surgery for any indication
  2. On cytotoxic chemotherapy for any indication (including methotrexate for arthritis)
  3. Hormonal therapy for cancer prevention (including tamoxifen). Note: treatment with finasteride/dutasteride for BPH does not render a participant ineligible
  4. Using medication which, in the opinion of the Investigator, would interfere with the study results (e.g., anti-inflammatory medications, antipsychotics, anticonvulsants with potential pain relief effects, immunomodulatory medications; blood thinners);
* Known sensitivity or allergy to grape powder;
* Nut allergies;
* Had received treatment for any type of internal cancer within 5 years prior to study entry;
* Had a history of or currently being treated for:

  1. Hepatitis;
  2. Diabetes (including insulin injections);
  3. Solid organ or bone marrow transplant
  4. Keloid formation
  5. Chronic renal or hepatic disorder
  6. Significant bleeding disorder
  7. Progressive neurodegenerative condition
  8. Swallowing disorder
* OTHER

  a. Any condition that might have compromised study results;
* Uncontrolled concurrent illness including ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, uncontrolled symptomatic cardiac arrhythmia, psychiatric illness/social situations that limited compliance with study requirements or other underlying serious medical condition which, in the investigator's opinion precluded study participation.

  b. Currently participating in any clinical testing; c. Received any investigational drug(s) within 28 days from Day 1.

Participants must also follow the following Subject Responsibilities:

Participants are not to consume the following foods during the study: Artichokes, figs, green tea, almonds, red fruits and vegetables, turmeric, olive oil, berries (blueberries, blackberries, grapes, raspberries, strawberries, goji berries, etc.), cocoa, dark chocolate, pomegranate, red wine

Participants are to limit the following foods during the study:

Coffee/Tea - 1X per day, beans/legumes - 2X per week, Soy foods (tofu, soy milk, miso, tempeh) 2X per week

Participants are not to consume the following supplements during the study: Multivitamin, Alpha lipoic acid, B vitamins, Coenzyme Q10, Elderberry, Ellagic acid, Fish oil, Flaxseed or flaxseed oil, Grapeseed extract, Green tea, Lycopene 6, Niacinamide, Quercetin, Resveratrol, Selenium, Turmeric, Vitamin C, E, K

Min Age: 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2025-09-09 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Biomarker - Myostatin | From start of enrollment to the end of treatment at 4 weeks
  Through serum analysis, myostatin will be measured in units of pg/mL at three points throughout the study.
Biomarker - IL-6 | From start of enrollment through treatment at week 4
  Through serum analysis, Interleukin-6 (IL-6) will be measured in units of pg/mL at three points throughout the study.
Biomarker - GDF-15 | From start of enrollment to the end of treatment at 4 weeks
  Through serum analysis, Growth Differentiation Factor 15 (GDF-15) will be measured in units of pg/mL at three points throughout the study.
BIomarker - BDNF | From start of enrollment through end of treatment at 4 weeks
  Through serum analysis, Brain-derived neurotrophic factor (BDNF) will be measured in units of pg/mL at three points throughout the study.
Biomarker - Cystatin C | From start of enrollment through the end of treatment at 4 weeks
  Through serum analysis, biomarker Cystatin C will be measured in units of pg/mL at three points throughout the study.
Biomarker - TNF-α | From start of enrollment through the end of treatment at 4 weeks
  Through serum analysis, biomarker Tumor necrosis factor-alpha will be measured in units of pg/mL at three points throughout the study.
Biomarker - CRP | From start of enrollment through the end of treatment at 4 weeks
  Through serum analysis, biomarker C-reactive protein (CRP) will be measured in units of pg/mL at three points throughout the study.
Biomarker - CCL-2/MCP-1 | From start of enrollment through the end of treatment at 4 weeks
  Through serum analysis, biomarker C-C motif chemokine ligand 2 / Monocyte chemoattractant protein 1 will be measured in units of pg/mL at three points throughout the study.
Biomarker - CAF | From start of enrollment through the end of treatment at 4 weeks
  Through serum analysis, biomarker C-terminal fragment of agrin (CAF) will be measured in units of pg/mL at three points throughout the study.
Biomarker - Malondialdehyde | From start of enrollment through the end of treatment at 4 weeks
  Through serum analysis, biomarker malondialdehyde will be measured in units of µM at three points throughout the study.

SECONDARY OUTCOMES:
Functional Cognition | From start of enrollment to the end of treatment at 4 weeks
  Montreal Cognitive Assessment (MoCA) - a brief cognitive screening tool that effectively detects mild cognitive impairment, offering greater sensitivity than other instruments like the MMSE. It assesses multiple cognitive domains and is validated for use in older populations.
Functional Muscle Strength - Bilateral Grip Strength | From start of enrollment to the end of treatment at 4 weeks
  Bilateral Grip Strength -Hydraulic Hand Dynamometer - a reliable indicator of overall muscular strength and has been correlated with functional status and health outcomes in older adults.
Functional Muscle Strength - Bilateral Pinch Strength | From start of enrollment to the end of treatment at 4 weeks
  Bilateral Pinch Strength -Hydraulic Pinch Gauge - provide insight into fine motor function and hand dexterity, which are crucial for daily activities.
Functional Muscle Strength - Standing Balance | From start of enrollment to the end of treatment at 4 weeks
  Standing Balance - Timed Up and Go (TUG) Test - a quick and effective measure of mobility and balance, predicting fall risk in older populations.
Functional Muscle Strength - Overall Physical Performance | From start of enrollment to the end of treatment at 4 weeks
  Overall Physical Performance - Short Physical Performance Battery (SPPB) -evaluates lower extremity function through balance, gait speed, and chair stand tests. It is a validated tool for assessing physical performance and predicting disability and mortality in older adults.
Functional Muscle Strength - Self-Reported Instrumental Activities of Daily Living | From start of enrollment to the end of treatment at 4 weeks
  Self-Reported Instrumental Activities of Daily Living - Lawton-Brody IADL Scale - assesses an individual's ability to perform complex daily tasks, providing insight into functional independence.
Body Composition Total Score | From start of enrollment to the end of treatment at 4 weeks
  A body composition total score is an indicator of an individual's overall health by quantifying their body's components (fat, muscle, bone, and water) and providing a numerical rating, often out of 100, that serves as a health risk indicator. A body composition analysis machine will be used for this calculation.

CONTACTS AND LOCATIONS:
Overall Officials: Brittany C Adams, Principal Investigator — Western New England University
Locations (1):
- Western New England University, Springfield, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Starting 6 months after publication
Access Criteria: Reasonable requests submitted to the corresponding author of any publications will be honored.

REFERENCES:
- [Background] Dautzenberg G, Lijmer J, Beekman A. Diagnostic accuracy of the Montreal Cognitive Assessment (MoCA) for cognitive screening in old age psychiatry: Determining cutoff scores in clinical practice. Avoiding spectrum bias caused by healthy controls. Int J Geriatr Psychiatry. 2020 Mar;35(3):261-269. doi: 10.1002/gps.5227. Epub 2019 Dec 27. PMID 31650623
- [Background] Graf C. The Lawton Instrumental Activities of Daily Living (IADL) Scale. Medsurg Nurs. 2009 Sep-Oct;18(5):315-6. No abstract available. PMID 19927971
- [Background] Phu S, Kirk B, Bani Hassan E, Vogrin S, Zanker J, Bernardo S, Duque G. The diagnostic value of the Short Physical Performance Battery for sarcopenia. BMC Geriatr. 2020 Jul 13;20(1):242. doi: 10.1186/s12877-020-01642-4. PMID 32660438
- [Background] Leger, H., Tittle, R., Dowdell, S., & Thompson, C., (2022). Comparison of the Validity of the Timed Up and Go Test (TUG) and Activities-specific Balance Confidence Questionnaire (ABC) to the 'Gold Standard' Berg Balance Scale (BBS) in Assessing Fall Risk in the Elderly Population. J Rehab Pract Res, 3(2):133. https://doi.org/10.33790/jrpr1100133
- [Background] MacDermid JC, Evenhuis W, Louzon M. Inter-instrument reliability of pinch strength scores. J Hand Ther. 2001 Jan-Mar;14(1):36-42. doi: 10.1016/s0894-1130(01)80023-5. PMID 11243558
- [Background] Reza MM, Subramaniyam N, Sim CM, Ge X, Sathiakumar D, McFarlane C, Sharma M, Kambadur R. Irisin is a pro-myogenic factor that induces skeletal muscle hypertrophy and rescues denervation-induced atrophy. Nat Commun. 2017 Oct 24;8(1):1104. doi: 10.1038/s41467-017-01131-0. PMID 29062100
- [Background] Nara H, Watanabe R. Anti-Inflammatory Effect of Muscle-Derived Interleukin-6 and Its Involvement in Lipid Metabolism. Int J Mol Sci. 2021 Sep 13;22(18):9889. doi: 10.3390/ijms22189889. PMID 34576053
- [Background] Kamper RS, Nygaard H, Praeger-Jahnsen L, Ekmann A, Ditlev SB, Schultz M, Hansen SK, Hansen P, Pressel E, Suetta C. GDF-15 is associated with sarcopenia and frailty in acutely admitted older medical patients. J Cachexia Sarcopenia Muscle. 2024 Aug;15(4):1549-1557. doi: 10.1002/jcsm.13513. Epub 2024 Jun 18. PMID 38890783
- [Background] Bagheri R, Rashidlamir A, Motevalli MS, Elliott BT, Mehrabani J, Wong A. Effects of upper-body, lower-body, or combined resistance training on the ratio of follistatin and myostatin in middle-aged men. Eur J Appl Physiol. 2019 Sep;119(9):1921-1931. doi: 10.1007/s00421-019-04180-z. Epub 2019 Jun 25. PMID 31240397
- [Background] Tabara Y, Kohara K, Okada Y, Ohyagi Y, Igase M. Creatinine-to-cystatin C ratio as a marker of skeletal muscle mass in older adults: J-SHIPP study. Clin Nutr. 2020 Jun;39(6):1857-1862. doi: 10.1016/j.clnu.2019.07.027. Epub 2019 Aug 6. PMID 31431305
- [Background] Renteria I, Garcia-Suarez PC, Fry AC, Moncada-Jimenez J, Machado-Parra JP, Antunes BM, Jimenez-Maldonado A. The Molecular Effects of BDNF Synthesis on Skeletal Muscle: A Mini-Review. Front Physiol. 2022 Jul 6;13:934714. doi: 10.3389/fphys.2022.934714. eCollection 2022. PMID 35874524
- [Background] Ladang A, Beaudart C, Reginster JY, Al-Daghri N, Bruyere O, Burlet N, Cesari M, Cherubini A, da Silva MC, Cooper C, Cruz-Jentoft AJ, Landi F, Laslop A, Maggi S, Mobasheri A, Ormarsdottir S, Radermecker R, Visser M, Yerro MCP, Rizzoli R, Cavalier E. Biochemical Markers of Musculoskeletal Health and Aging to be Assessed in Clinical Trials of Drugs Aiming at the Treatment of Sarcopenia: Consensus Paper from an Expert Group Meeting Organized by the European Society for Clinical and Economic Aspects of Osteoporosis, Osteoarthritis and Musculoskeletal Diseases (ESCEO) and the Centre Academique de Recherche et d'Experimentation en Sante (CARES SPRL), Under the Auspices of the World Health Organization Collaborating Center for the Epidemiology of Musculoskeletal Conditions and Aging. Calcif Tissue Int. 2023 Feb;112(2):197-217. doi: 10.1007/s00223-022-01054-z. Epub 2023 Jan 12. PMID 36633611
- [Background] Rosner B. Fundamentals of Biostatistics. 7th ed. Boston, MA: Brooks/Cole; 2011.
- [Background] von Haehling S, Morley JE, Anker SD. An overview of sarcopenia: facts and numbers on prevalence and clinical impact. J Cachexia Sarcopenia Muscle. 2010 Dec;1(2):129-133. doi: 10.1007/s13539-010-0014-2. Epub 2010 Dec 17. PMID 21475695
- [Background] Maher, P. Grapes and the Brain. In Grapes and Health; Pezzuto, J.M., Ed.; Springer International Publishing: Cham, Switzerland, 2016; pp. 139-161.
- [Background] Pezzuto JM. Grapes and human health: a perspective. J Agric Food Chem. 2008 Aug 27;56(16):6777-84. doi: 10.1021/jf800898p. Epub 2008 Jul 29. PMID 18662007